CLINICAL TRIAL: NCT03514199
Title: Mediterranean-type Diet for Older Adults With Obstructive Sleep Apnea: Randomized Clinical Trial - MedOOSA Project
Brief Title: Mediterranean-type Diet for Older Adults With Obstructive Sleep Apnea
Acronym: MedOOSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 79655917700005327
Record Dates: First submitted 2018-04-20; First posted 2018-05-02 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-02

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial will be conducted and the sample will consist of 50 participants who performed portable respiratory polysomnography. Cases with AHI between 15 and 50 events per hour will be sent for medical evaluation to identify inclusion/exclusion criteria. Eligible individuals who agree to participate in the study, after signing the Informed Consent Term, will perform physical, biochemical, questionnaire and randomized to receive guidelines on the Mediterranean-type diet or low-fat diet.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean-type diet (Experimental): Recommends high consumption of whole grains, vegetables, nuts, fruits, vegetables and olive oil as the main source of fat used for salads. Moderate to high fish consumption and low consumption of red and processed meats. Poultry and dairy products (such as yogurt or cheese) will be consumed in small quantities and moderate consumption of alcohol, usually in the form of red wine, will be recommended with meals for usual drinkers.
  Interventions: Other: Mediterranean-type diet
- Low fat diet (Active Comparator): It recommends reducing the intake of foods rich in fats, especially those saturated and hydrogenated.
  Interventions: Other: Low fat diet

INTERVENTIONS:
Other: Mediterranean-type diet — Recommendations: ingest whole grains; three or more servings/day (various fresh fruits/vegetables); three or more servings/week of fish or seafood; white meat to red and processed meat (red meat to one serving or less/day); oilseed mix - 30g/day (nuts: 15g/day, almonds: 7.5g/day, hazelnuts: 7.5g/day); extra virgin olive oil (30ml/day: 2 soup spoons/day) as the main source of fat in the salads; two or more servings per week of "sofrito"; two servings/day of low-fat dairy products; limit to one serving/week the intake of fatty and cured cheeses; recommendation of 7 glasses per week of red wine (recommendation for habitual drinkers): 1 cup/day of 100ml for women and 1-2 cups/day of 150ml for men; limit to one serving/week the intake of chocolate with more than 50% cocoa.
  Arms: Mediterranean-type diet
Other: Low fat diet — Recommendations: choose grilled, cooked, baked or soaked preparations; avoid frying (sweet or salty); avoid excess fat in the preparations and season the foods with herbs at will (marjoram, basil, oregano, onion, green seasoning, sweet pepper, sage, etc.); avoid frequent ingestion of sausages such as ham, turkey breast, among others; avoid eating fatty meats and strip the skin of poultry before preparation; avoid eating sweets and fatty foods; avoid ingesting bakery products, such as leafy, tart, savory pasta.
  Arms: Low fat diet

SUMMARY:
The majority of the elderly present with sleep apnea and mortality is significantly higher in this group. Sleep apnea runs the risk of developing diseases, especially hypertension and cardiovascular disease, while the Mediterranean diet is associated with reduced risk.

No study evaluated the effect of the Mediterranean diet on the apnea and hypopnea index in the elderly. Therefore, the present work intends to evaluate the effect of the intervention with the Mediterranean diet on the apnea-hypopnea index in the elderly with moderate sleep apnea.

The hypothesis study is that the elderly with moderately severe sleep apnea under a Mediterranean-type diet will modify AHI in the short term, regardless of weight change, due to changes in body volume and ingestion, especially those related to body water.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To evaluate the effect of the Mediterranean diet intervention on the apnea-hypopnea index in the elderly with moderate-severe sleep apnea.

SECONDARY OBJECTIVES:

* To compare the effect of intervention with Mediterranean diet on the effect of low-fat diet (control) on anthropometric variables (BMI, neck and waist circumferences) and bioimpedance (body water, lean mass, fat mass).
* To compare the effect of the intervention with a diet of the Mediterranean type to the effect of the intervention with a low-fat diet (control) on glycolipid profile, C-reactive protein, Sodium, and Potassium.
* To compare the effect of the Mediterranean diet intervention on the effect of the low-fat diet (control) on blood pressure: systolic, diastolic and heart rate measured in 24-hour ABPM.

PROCEDURES:

All variables will be measured equally in the two groups: Mediterranean diet and control diet. The provision of extra virgin olive oil and oilseeds will be provided free to participants randomized to the Mediterranean diet at visits 1 and 2 and participants randomized to the control diet will receive nutritional guidelines. There will be no caloric restriction for both groups, nor will there be any increase in physical activity.

All participants will be interviewed by a nutritionist and a nutritionist at the baseline and at all subsequent visits, and the dietary guidelines will be given by the same nutritionist. Evaluations with participants from both groups will be organized separately for each of the groups. All participants will be instructed not to use multivitamins or antioxidant supplements during the study period.

ASSESSMENT OF ADHERENCE TO THE MEDITERRANEAN DIET:

A questionnaire with 14 items (Annex 3) assessing adherence to the Mediterranean diet will be used. A value of 0 (not compatible) or 1 (compatible) will be assigned to each item answered on the diet. Higher scores will reflect better adherence to the diet. High adherence will be set when matching at least 11 of the 14 items.

RANDOMIZATION:

The randomization to the diet group of the Mediterranean type or Diet Control will be performed by withdrawing the envelope in groups of 4 following random numbers generated by computer.

SAMPLE SIZE The sample size calculation is based on the study "Effect of Mediterranean diet versus prudent diet combined with physical activity on OSAS: a randomized trial" 45. For a 5% alpha error and 80% power, the calculated sample size was 24 patients in each group to detect an effect size of 0.25 standard deviation. However, considering withdrawals, withdrawal of consent, absenteeism, and case losses during the study period, up to 25 patients will be evaluated in the Mediterranean diet group and 25 in the control diet group.

STATISTICAL ANALYSIS The demographic characteristics and other variables of interest of the participants of the Mediterranean diet and Diet control groups will be compared using the Student's t-test or the chi-square test. Paired t-test or non-parametric test will be performed to compare measures at baseline and after two months of intervention within each group. Differences of measures of interest will be determined between the groups using covariance analysis (ANCOVA) controlled by the corresponding baseline levels, sex, and age or by non-parametric test. The transformation to log for data that is not normally distributed will be used. The significance of P <0.05 will be considered significant. The analyzes will be performed with the IBM SPSS Statistics version 20 program.

ELIGIBILITY:
Inclusion Criteria:

* Agreement to sign the ICF;
* AHI between 15 and 50 events/h;
* Age between 65 and 80 years;
* Both sexes;
* BMI between 27-39.9 kg / m2.

Exclusion Criteria:

* In treatment for sleep apnea;
* Predominantly central sleep apnea;
* Feed predominantly of meals provided by third parties;
* Gastrointestinal disease, with intolerance to fat intake;
* Impossibility to follow the Mediterranean diet due to the presence of mastication and/or swallowing disorders;
* History of food allergy with hypersensitivity to any of the components of olive oil and/or oleaginous;
* Eating habits in the last two months that characterize the diet of the Mediterranean;
* Significant alterations in appetite in the last three months or change of weight over 5 kg in the last three months;
* Illegal use of drugs or chronic alcoholism, clinically significant depression or ongoing psychiatric care;
* Inability to communicate;
* Severe chronic diseases;
* Self-reported terminal disease;
* Plan to move city in two months;
* Participation in another clinical trial.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Apnea-hypopnea index | 12 weeks
  Evaluated with portable polygraphy.

SECONDARY OUTCOMES:
Body weight | 12 weeks
  Clinical scale will be used with 100g precision.
Body composition | 12 weeks
  Measured by bio-impedance. The device used will be Biodynamics®, model 450, version 5.1 International.
glucose | 12 weeks
  Blood collection will be performed between 07:30 and 9:30 a.m. in the morning of 12 hours, by a trained technician who will obtain a blood sample by venipuncture.
Cholesterol total | 12 weeks
  Blood collection will be performed between 07:30 and 9:30 a.m. in the morning of 12 hours, by a trained technician who will obtain a blood sample by venipuncture.
LDL-Cholesterol | 12 weeks
  Blood collection will be performed between 07:30 and 9:30 a.m. in the morning of 12 hours, by a trained technician who will obtain a blood sample by venipuncture.
HDL-cholesterol | 12 weeks
  Blood collection will be performed between 07:30 and 9:30 a.m. in the morning of 12 hours, by a trained technician who will obtain a blood sample by venipuncture.
Triglycerides | 12 weeks
  Blood collection will be performed between 07:30 and 9:30 a.m. in the morning of 12 hours, by a trained technician who will obtain a blood sample by venipuncture.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Martinez, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre

IPD SHARING:
Plan to Share IPD: Undecided